CLINICAL TRIAL: NCT06181955
Title: Effectiveness of Extracorporeal Shock Wave Therapy on Improving Functional Ability in Knee Osteoarthritis (Grade iv)
Brief Title: Extracorporeal Shock Wave Therapy in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AWH/EC/03/2021/2
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Physical therapy; Lower Extremity Functional Scale score; Ultrasound therapy; Exercises; Quadriceps
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Two group experimental-control design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The participants in this group received Extracorporeal Shock Wave Therapy (ESWT) in addition to conventional physical therapy.
  Interventions: Other: Extracorporeal Shock Wave Therapy; Other: conventional physical therapy
- Control group (Active Comparator): The participants in this group received conventional physical therapy only.
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: Extracorporeal Shock Wave Therapy — The ESWT was performed by an ESWT instrument (Chattanooga) once a week for four consecutive weeks (a total of four sessions).
  Arms: Experimental
Other: conventional physical therapy — Conventional physical therapy consisted of ultrasound therapy and three types of knee-strengthening exercises.

SUMMARY:
The present study has examined the effectiveness of extracorporeal shock wave therapy along with conventional physical therapy on functional ability in grade IV knee osteoarthritis. Intervention program was performed for four weeks. Conventional physical therapy included ultrasound therapy, isometric quadriceps, straight leg raising (SLR) and isometric hip adductor strengthening exercises. Functional ability was assessed using the Lower Extremity Functional Scale (LEFS) score.

ELIGIBILITY:
Inclusion Criteria:

* Grade IV primary knee Osteoarthritis (OA) diagnosed by an orthopaedic surgeon based on the Kellgren-Lawrence score

Exclusion Criteria:

* Secondary knee OA,
* rheumatoid arthritis,
* psoriatic arthritis,
* the presence of any red flags (metastatic growth, thrombophlebitis),
* neurologic or psychiatric impairments,
* tissue injuries of the knee joint,
* previous knee joint replacement or other surgeries in the knee joint,
* already received ESWT,
* Intra articular injection
* unable to walk independently

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Functional Scale (LEFS) score | 4 weeks
  It is a measurement tool used to assess the functional status and ability of individuals with lower extremity musculoskeletal conditions or injuries. The LEFS consists of 20 items and each item is rated on a scale from 0 to 4, with 0 indicating extreme difficulty to perform the activity and 4 indicating no difficulty at all. The scores for all items are summed to obtain a total score ranging from 0 to 80.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, MPTh, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No